CLINICAL TRIAL: NCT07105969
Title: Evaluation Stability the Antibacterial Efficacy and of Strontium Incorporated Hydroxyapatite [Sr-HA] Coated Mini-screws Used for Maxillary Canine Retraction: A Randomized Clinical Trial
Brief Title: Strontium-Hydroxyapatite Coated Mini-Screws: Antibacterial Effect and Stability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS.25.04.20
Record Dates: First submitted 2025-06-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gingival Inflammation and Loss the Orthodontic Mini-screws
Keywords: ▪️Sr-HA ▪️Mini-screw stability ▪️Antibacterial afficacy
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : uncoated OMSs. (No Intervention): Mini- screw uncoated by Sr-HA
- Group 2: coated OMSs by Sr-HA (Experimental): Mini-screw coated by Sr-HA
  Interventions: Other: Strontium Incorporated Hydroxyapatite [Sr-HA] coated mini-screws purchased from Dentarum company

INTERVENTIONS:
Other: Strontium Incorporated Hydroxyapatite [Sr-HA] coated mini-screws purchased from Dentarum company — Maxillary canine retraction by mini-screw loaded with 150g Niti coil spring
  Other Names: Mini -screw stability
  Arms: Group 2: coated OMSs by Sr-HA

SUMMARY:
This randomized controlled clinical trial aims to evaluate the antibacterial efficacy and stability of strontium-incorporated hydroxyapatite (Sr-HA) coated orthodontic mini-screws (OMSs) used for maxillary canine retraction. A double-blind, split-mouth design was employed, involving 20 patients (aged 16-20 years), each receiving two titanium alloy mini-screws (1.6 mm × 8 mm): one coated with Sr-HA (5% concentration via electrochemical deposition) and one uncoated control. A total of 40 mini-screws were assessed. Following upper first premolar extractions, canine retraction was initiated using 150 g NiTi coil springs on 17×25 SS archwires. Mini-screws were placed between the upper second premolar and first molar without flap elevation or pilot hole drilling. Parameters including screw stability, antimicrobial activity, and gingival blood flow were monitored over a 4-month period. The incorporation of Sr-HA is hypothesized to enhance mini-screw osseointegration, reduce peri-implant inflammation, and improve clinical outcomes by leveraging the osteogenic and antibacterial properties of strontium. This study aims to provide evidence supporting the use of Sr-HA coatings to reduce mini-screw failure rates in orthodontic treatment.

DETAILED DESCRIPTION:
Aim of the study:

The aim of this study is to evaluate the antibacterial efficacy and stability of strontium- incorporated hydroxyapatite (Sr-HA) coated orthodontic mini- screws used in maxillary canine retraction in comparison to uncoated mini- screws.

Material and methods:

1. All patients will be treatment with fixed appliance and Roth type brackets where leveling and alignment will be done utilizing nickel titanium.
2. Extraction the upper first premolars and retraction the canine will be done using 17 ×25 SS wire.
3. A periapical X-ray will be taken to confirm the mini screw position to avoid interference with adjacent root and to ensure that there are no periapical lesion.
4. Symmetrical orthodontic miniscrews will be inserted between the second premolar and first molar.
5. The OMSs that will be used in this study will be self-drilling, conical in shape, 1.6 mm in diameter, and 8 mm in length, constructed of titanium alloy, i well be purchased from Dentaurum company [Germany].
6. The orthodontic main screws were loaded with a 150 g NiTi coil spring.
7. On one side, a coated will be inserted, and on the other side, an uncoated will be used for the same patient.
8. Coated materials will utilize [Strontium incorporated hydroxyapatite] applied by electrochemical deposition and concentration percentage about 5 % .
9. No mucoperiosteal flap will be raised, and no pilot hole will be made during the procedure.
10. Will be assessed throughout follow-up periods of up to four months.

Outcome Measurement:

1. Assessment Orthodontic mini-screws stability (coated and uncoated) using Periotest device .
2. Evaluate antimicrobial effect of Strontium incorporated Hydroxyapatite using Enzem- Linked Immunosorbent technique .
3. Evaluate blood flow by periodental probe.
4. Gingival health by visual assessment .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients within an age range (16-20) years.
2. Orthodontic treatment plan requiring the extraction of the upper first premolars.
3. Patients have fully permanent teeth are erupted (third molars are not included).
4. No previous orthodontic treatment
5. No medical problem that could interfere with treatment.

Exclusion Criteria:

1. Presence of problematic healing such as, compromised immune defense, bleeding disorder, pathological bone quality, and xerostomia.
2. Inadequate oral hygiene.
3. Heavy smoking

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Orthodontic mini-screws stability | Four mounth
  Mean value of orthodontic mini-screw stability assessed using the Periotest device
  Measurement Tool: A Periotest device (manufactured by Medizintechnik Gulden, Germany) will be used to evaluate the mechanical stability of the orthodontic mini-screws.
  Unit of Measure: Periotest Values (PTV), expressed as numerical values ranging from -8 (high stability) to +50 (low stability).
  Assessment Method: The stability of both coated (Strontium-incorporated Hydroxyapatite) and uncoated orthodontic mini-screws will be measured and compared at specific time intervals throughout the study period.

SECONDARY OUTCOMES:
Anti microbial effect | Four mounth
  Mean concentration of bacterial adhesion on orthodontic mini-screw surfaces assessed by Enzyme-Linked Immunosorbent Assay
  Measurement Tool: Enzyme-Linked Immunosorbent Assay (ELISA) will be employed to quantify the level of bacterial colonization on the surface of the mini-screws.
  Unit of Measure: Colony Forming Units per milliliter (CFU/mL), or Optical Density (OD) values at a specific wavelength (typically 600 nm), depending on the ELISA protocol used.
  Assessment Method: The antimicrobial effect of the Strontium-incorporated Hydroxyapatite coating will be evaluated by comparing the level of bacterial adhesion on coated versus uncoated mini-screw surfaces.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
individual participants available upon request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT07105969/Prot_SAP_001.pdf